CLINICAL TRIAL: NCT04582058
Title: Mobile Health of Lifestyle to Patients With Cardiac Electronic Implantable Device: Randomized Clinical Trial
Brief Title: Mobile Health For Pacemaker Patientes
Acronym: MHOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InCor Heart Institute (Other)
Collaborators: Spectator Healthcare Technology (Unknown)
Responsible Party: Principal Investigator, Martino Martinelli Filho, MD, PHD, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHOL
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Sedentary Behavior; Anxiety Disorders; Depressive Disorder; Quality of Life
Keywords: cardiovascular disease; Mobile Health
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior; Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Interventional Group (IG): Mobile Health to patients with an orientation about daily activities and protocol of physical exercise Control Group (CG): normally follow up, without mobile health
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): Control Group (CG): Standard of care, normally follow up, without mobile health
- Interventional Group (IG) (Experimental): Interventional Group (IG): Mobile Health to patients with an orientation about daily activities and protocol of physical exercise
  Interventions: Behavioral: Mobile Health of lifestyle

INTERVENTIONS:
Behavioral: Mobile Health of lifestyle — Mobile health of lifestyle with an orientation about daily activities and necessary care to patients with CEID, and protocol of exercise training with images and guidelines to execute five days per week, with a duration of 50 minutes, and space for doubts which patients could send message to researcher.
  Arms: Interventional Group (IG)

SUMMARY:
Previous studies suggested that most patients with Cardiac Electronic Implantable devices have a perception of describing the lifestyle due to a limitation of daily activities and physical exercise, besides the consequences in the psychological aspects such as anxiety and depression. The MHOL-CEID is a randomized controlled trial that Verifies the effectiveness of the Mobile Health of lifestyle that focuses on aspects of physical functional, psychosocial, and quality of life of patients with Cardiac Electronic Implantable Device.

DETAILED DESCRIPTION:
Cardiovascular diseases represent one of the main causes of death in the Brazilian population, as well as dysfunctions of the heart conduction system. In an attempt to treat and correct heart conduction system dysfunctions, Cardiac Electronic Implantable Device (CEID) was developed. Most people with CEID have a perception of describing the lifestyle due to a limitation of daily activities and physical exercise, besides the consequences in the psychological aspects such as anxiety and depression. These changes in the psychosocial conduct of patients with CEID are due to the lack of knowledge and the lack of effective guidance, being of fundamental importance to elaborate the resources of education in health for patients with CEID. Health promotion through educational intervention is a recognized strategy and an Internet approach to the mobile health proposal is a recognized and promising practice.

This randomized controlled study is been conducted to verify the effectiveness of the Mobile Health of lifestyle that focuses on aspects of physical functional, psychosocial, and quality of life of patients with CEID. The hypothesis is that the use of Mobile Health of lifestyle provides greater physical functional, psychological aspects, and quality of life to patients with CIED.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to randomization and any study procedure;
* Patients with any CIED
* Access to the internet
* Clinical stability in the last 3 weeks
* With left ventricular ejection fraction (LVEF) greater than 40%
* Skill to conduct the self-monitoring of intensity in physical activity
* New York Heart Association classification 1 or 2

Exclusion Criteria:

* Unstable angina
* Uncontrolled systemic arterial hypertension
* Cardiac arrhythmia effort- induced
* People with a musculoskeletal or neurological problem
* Cognitive disability
* Patients opposed to the participation in the research
* Other concomitants cardiovascular disease, including uncontrolled diabetes mellitus (systemic hypertension without target-organ impairment is allowed);
* Moderate or severe chronic obstructive pulmonary disease;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-11-20 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | Six minutes
  Six walk minutes test to assess and measures the distance that patient can walk on a flat in a period of 6 minutes

SECONDARY OUTCOMES:
Quality of life of patients | Thirty minutes
  SF 36 questionnaire, evaluate health-related quality of life. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH).
Anxiety and depression | Thirty minutes
  Hospital anxiety and depression scale, which consist 14 questions that evaluate how patients felt during the previous week. Scores with range 0-21.
Level of physical activity | Thirty minutes
  IPAQ questionnaire, • To assesses the types of intensity of physical activity and sitting time that patients do on daily lives activities, and are considered to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Martino MM Martinelli Filho, PHD, Principal Investigator — InCor Heart Institute
Locations (1):
- Martino Martinelli Filho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided